CLINICAL TRIAL: NCT04733404
Title: A Prospective, Multicenter, Objective Performance Criteria Study to Evaluate the Safety and Effectiveness of Dragonfly Transcatheter Mitral Valve Repair System for the Treatment of Functional Mitral Regurgitation (FMR) Subjects.
Brief Title: Safety and Effectiveness Study of Dragonfly System for Functional Mitral Regurgitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DragonFly-02
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-06

CONDITIONS: Mitral Regurgitation Functional

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dragonfly Mitral Valve Repair System (Experimental): The experimental group is allocated to use a novel mitral valve repair system for edge-to-edge repair manufactured by Hangzhou Valgen Medtech Co., Ltd.
  Interventions: Device: Dragonfly Transcatheter Mitral Valve Repair System

INTERVENTIONS:
Device: Dragonfly Transcatheter Mitral Valve Repair System — To conduct edge-to-edge repair with Dragonfly System under the guidance of transesophageal echocardiography.

SUMMARY:
To confirm the effectiveness and safety of the Dragonfly transcatheter mitral valve repair system for the treatment of chronic moderate to severe (3+) or severe (4+) functional mitral regurgitation (FMR) who remained clinically symptomatic after guideline-directed medical treatment.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, objective performance criteria design. Patients are chronic moderate to severe (3+) or severe (4+) functional mitral regurgitation (FMR) who remained clinically symptomatic after guideline-directed medical treatment. After signing an informed consent form, subjects are enrolled and treated with the DragonFly Transcatheter Mitral Valve Repair System. All subjects receive clinical follow-up immediately after procedure, before discharge, 30 days after procedure, 6 months after procedure, and 12 months after procedure.

The primary outcome is defined as a composite measure include all-cause mortality and recurrent heart failure hospitalization at 12 months after procedure.

The secondary outcomes include acute procedural success, acute device success, mitral regurgitation degree (MR≤2+), recurrent heart failure hospitalization, NYHA class I or II at 30 days, 6 months, and 12 months, and the improvement in 6 minutes walk test distance, left ventricular end-diastolic volume, quality of life change as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) score from baseline at 12 months after procedure.

The safety endpoints include major adverse events (MAEs) at 30 days and 12 months after procedure, and all-cause mortality, cardiac mortality at 30 days, 6 months, and 12 months after procedure.

To evaluate the safety and effectiveness of the Valgen Medtech DragonFly Transcatheter Mitral Valve Repair System in the treatment of patients with chronic moderate to severe (3+) or severe (4+) functional mitral regurgitation (FMR) who remained clinically symptomatic after guideline-directed medical treatment, and to evaluate the product performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 yrs.
2. Symptomatic functional mitral regurgitation (FMR) (≥3+) due to ischemic or non-ischemic cardiomyopathy Note 1: Functional MR requires the presence of overall or localized LV wall motion abnormalities that are considered to be the primary cause of MR. Despite the eligibility, subjects may not enroll if leaflet prolapse or other evidence of degenerative MR is present.

   Note 2: An Eligible transthoracic echocardiography must be obtained at least 30 days after the subject has been stabilized on optimal therapy with Guideline Directed Medical Therapy (GDMT), and after meeting two of the following conditions:
   1. GDMT dose increase of no greater than 100% or decrease of no greater than 50%.
   2. Coronary revascularization and/or implantation of a cardiac resynchronization therapy device (CRT or CRT-D) or reprogramming of the implanted CRT or CRT-D resulting in an increase in biventricular pacing (from <92% to ≥92%).
3. Subjects have been adequately treated according to applicable criteria, including treatment for coronary artery disease, left ventricular dysfunction, mitral regurgitation, and heart failure (e.g., with cardiac resynchronization therapy (CRT or CRT-D), coronary revascularization, and/or have received stable GDMT, as defined in (Appendix IV: Definition of GDMT), confirmed by the local heart team.
4. NYHA functional class II to IVa.
5. Left ventricular ejection fraction (LVEF) ≥ 20% and ≤50%.
6. Left ventricular end-systolic dimension (LVESD) ≤ 70 mm.
7. Anatomically suitable for transcatheter mitral valve repair by edge-to-edge technique and can be treated by the DragonflyTM device.
8. Elevated BNP >150 pg/ml or corrected NT-proBNP ≥600 pg/ml or heart failure hospitalization within the past 12 months ('corrected' refers to a 4% reduction in the BNP or NT-proBNP cutoff for every increase of 1 kg/m2 in BMI above a reference BMI of 20 kg/m2).
9. Transseptal catheterization and femoral vein access is determined to be feasible.
10. The subject or subject's legal representative has been informed of the nature of the trial, willing to accept the experimental tests, and has provided written informed consent.

Exclusion Criteria:

1. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
2. The presence of other severe heart valve disease requiring surgical intervention.
3. Prior mitral valve leaflet surgery or transcatheter mitral valve intervention.
4. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, infiltrative cardiomyopathy (e.g., amyloidosis, hemochromatosis, sarcoidosis, etc.), or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology.
5. Moderate to severe right heart dysfunction or an estimated pulmonary artery systolic pressure (PASP) > 70 mmHg assessed by echocardiography.
6. History of acute myocardial infarction in the prior 4 weeks or untreated clinically significant coronary artery disease requiring revascularization.
7. Any percutaneous cardiac intervention within the 30 days, or any cardiac surgery within the 6 months prior to randomization, or any implant of any Cardiac Resynchronization Therapy (CRT) or Cardiac Resynchronization Therapy with cardioverter-defibrillator (CRT-D) or Implantable Cardioverter Defibrillator (ICD) within the last 30days prior to subject registration.
8. In the judgment of the investigator, the subject's femoral vein is unable to accommodate a 25F catheter or has an ipsilateral deep venous thrombosis; or the anatomy is not accessible for transseptal puncture.
9. Subjects in whom transesophageal echocardiography (TEE) or general anesthesia is contraindicated.
10. End-stage heart failure (ACC/AHA stage D), or prior orthotopic heart transplantation, or on the waiting list for heart transplantation.
11. Active endocarditis, or active rheumatic heart disease, or leaflets degenerated from either endocarditis or rheumatic disease.
12. Severe Chronic Obstructive Pulmonary Disease (COPD) (requiring continuous home oxygen therapy or long-term application of steroid hormone medication).
13. Cerebrovascular accident within 30 days prior to randomization or symptomatic severe carotid stenosis (> 70% by ultrasound), or carotid artery stenting within 30 days.
14. Evidence of acute peptic ulcer or gastrointestinal hemorrhage in the prior 3 months.
15. Hemorrhagic or coagulopathic disorders, contraindications to antithrombotic medication.
16. Modified Rankin Scale ≥4.
17. The subjects suffer from diseases that may lead to difficulty in evaluating treatment (e.g., cancer, severe metabolic disease, psychosis, etc.).
18. Pregnant or breastfeeding women, or women who plan to become pregnant within the next 12 months. Note: Women of childbearing age should take a pregnancy test with a negative result within 14 days prior to registration and use scientifically safe contraception
19. Hemodynamic instability defined as systolic pressure < 90 mmHg without afterload reduction, cardiogenic shock, or the need for inotropic support or an intra-aortic balloon pump.
20. Active infections requiring antibiotic therapy (in the case of temporary illness, antibiotics must be discontinued for at least 14 days before the subject can be enrolled).
21. Currently participating in an investigational drug or another device study that has not completed its primary endpoints or would clinically interfere with the endpoint of this study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
22. In the judgment of the investigator, subjects may not complete the trial according to poor compliance or in other circumstances when the investigator determines that the subject is unfit to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-12 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with composite measures- All-cause death and recurrent HF hospitalizations. | 12 months
  A composite of all-cause death or recurrent heart failure (HF) hospitalizations.

SECONDARY OUTCOMES:
Mitral regurgitation severity | 30 days, 6 months, 12 months
  Percentage of patients with mitral regurgitation of 2+ or less.
Recurrent heart failure (HF) hospitalizations | 30 days, 6 months, 12 months
  Number of patients with incidence of re-hospitalizations for heart failure after Dragonfly implantation.
NYHA Class | 30 days, 6 months, and 12 months
  Number of patients with New York Heart Association (NYHA) Function Class I or II.
Change in 6 minutes walk test distance | 12 months
  Improvement in 6 Minute Walk Test distance at 12 months over baseline.
Quality of life improvement | 12 months
  Improvement in quality of life (QoL) at 12 months over baseline, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).
Left Ventricular End Diastolic Volume (LVEDV) | 12 months
  Left Ventricular End Diastolic Volume (LVEDV) as determined by the core echocardiography laboratory from a transthoracic echocardiogram (TTE).
Acute procedural success | Immediately after procedure, Discharge: The day after the patient's exit from the cardiac catheterization laboratory
  Successful in Dragonfly implantation, and residual MR of 2+ or less at discharge. An echocardiography echocardiogram at 30 days can be accepted if the discharge image was not available or hard to interpret. A death before discharge or a re-operation of mitral valve prior to 30 days is defined as acute procedure failure.
Acute device success | Immediately after procedure
  One or more Dragonfly devices are successfully delivered and released, edge-to-edge leaflet repair confirmed by echocardiogram, and successfully withdrawal of the delivery catheter.

OTHER OUTCOMES:
Incidence of major adverse events (MAEs) | 30 days, and 12 months
  MAE is defined as a combined clinical endpoint of death, stroke, myocardial infarction, renal failure, and nonelective cardiovascular surgery for device or procedure-related adverse events occurring after transseptal catheterization.
All-cause mortality | 30 days, 6 months, and 12 months
  Percentage of all-cause death includes cardiac death, non-cardiac death, and death from unknown causes.
Cardiac mortality | 30 days, 6 months, and 12 months
  Percentage of cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, MD, PH.D, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No